CLINICAL TRIAL: NCT04741659
Title: Tidal Volume in Patients With "de Novo" Acute Hypoxemic Respiratory Failure Receiving Non-invasive Respiratory Supports: a Pilot Study
Brief Title: Tidal Volume in Patients With "de Novo" Acute Hypoxemic Respiratory Failure
Acronym: DENOVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Stefano Nava, Professor of Respiratory Medicine/ Alma Mater Studiorum University of Bologna (IT)- Director of Respiratory and Critical Care Unit/ S.Orsola-Malpighi University Hospital, Bologna (IT), IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 691/2020/Sper/AOUBo
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: De novo; ARF
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- spontaneous breathing trial (Placebo Comparator): the patients will be asked to breathe spontaneously using their actual low oxygen flow
  Interventions: Device: Ventimask; Device: High Flow Nasal cannula (HFNC); Device: Helmet CPAP; Device: Non Invasive Ventilation (NIV)
- High Flow Nasal cannula (HFNC) (Active Comparator): The patients will be asked to breathe with HFNC of 40 L/min
  Interventions: Device: Ventimask; Device: High Flow Nasal cannula (HFNC); Device: Helmet CPAP; Device: Non Invasive Ventilation (NIV)
- Helmet CPAP (Active Comparator): the patients will be asked to breathe with the Helmet CPAP
  Interventions: Device: Ventimask; Device: High Flow Nasal cannula (HFNC); Device: Helmet CPAP; Device: Non Invasive Ventilation (NIV)
- Non Invasive Ventilation (NIV) (Active Comparator): the patients will be asked to breathe with the support of a ventilator via a oro-nasal interface
  Interventions: Device: Ventimask; Device: High Flow Nasal cannula (HFNC); Device: Helmet CPAP; Device: Non Invasive Ventilation (NIV)

INTERVENTIONS:
Device: Ventimask — The patients will be asked to breathe spontaneously using their actual low oxygen flow
Device: High Flow Nasal cannula (HFNC) — The patients will be asked to breathe using high flow nasal cannula (HFNC). Air flow will set up to 60 l/m, temperature according to patient's comfort and FiO2 in order to obtain SpO2 values >/= 92%
Device: Helmet CPAP — The patients will be asked to breathe with Helmet. CPAP will set at 10 cmH2O and FiO2 in order to obtain SpO2 values >/= 92%
Device: Non Invasive Ventilation (NIV) — the patients will be asked to breathe with the support of a ventilator via a oro-nasal interface

SUMMARY:
Protective ventilation can be difficult to achieve during noninvasive ventilation for "de novo"acute hypoxemic respiratory failure (i.e., not due to exacerbation of chronic lung disease or cardiac failure).Recent data suggest patient self-inflicted lung injury (P-SILI) as a possible mechanism aggravating lung damage in these patients.

The aim of this study is evaluate the tidal volume, measured by respiratory inductance plethysmography, in patients receiving different non invasive respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* Acute Respiratory Failure (ARF) ( 100 <PaO2/FiO2 <300) due to Covid-19 infection
* Informed consent
* Enrollment within the first 24 hours after ARF

Exclusion Criteria:

* Clinical, radiological or istological evidence of chronic pulmonary disease.
* Body Mass Index (BMI) > 30 kg/m2;
* Previous diagnosis of Obstructive sleep apnea syndrome (OSAS)
* Chest wall disease
* Heart failure
* Severe hemodynamic instability ( need for amine support)
* Acute coronary syndrome (ACS)
* Severe arrhythmia
* Patients unable to protect respiratory airways
* Respiratory arrest and need for endotracheal intubation
* Pregnancy
* Need for sedation
* Home long-term oxygen therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
respiratory pattern | 30 minutes
  the way the patient is breathing recorded by respiratory inductance plethysmography (RIP)
respiratory mechanics | 30 minutes
  the inspiratory effort of the patient recorded by esophageal pressure

SECONDARY OUTCOMES:
changes in Arterial Blood Gases (ABGs) | immediately after intervention
  Arterial Blood Gases, namely arterial oxygen (PaO2) and carbon dioxyde (PaCO2) tension will be analyzed from a sample taken from the arterial artery
Dyspnea score | immediately after intervention
  Dyspnea will be recorded using the Borg scale that is a numeric scale where 0 is no dyspnea and 10 the maximal dyspnea that a patient can imagine
Comfort score | immediately after intervention
  this will be assessed using a dedicated visual analog scale (VAS with a length of 20 cm)
Blood pressure (BP) and Heart rate (HR) measurements | 30 minutes
  blood pressure and heart rate will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, MD, Principal Investigator — Alma Mater Studiorum University of Bologna (IT)- Director of Respiratory and Critical Care Unit/ IRCSS S.Orsola-Malpighi University Hospital, Bologna (IT)
Locations (1):
- IRCCS Policlinico di Sant'Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No